CLINICAL TRIAL: NCT02099019
Title: Usefulness of Coronary Computed Tomography Angiography for Therapeutic Decision- Making; Revascularization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2013-0084
Record Dates: First submitted 2014-03-19; First posted 2014-03-28 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease, Ischemic Heart Disease
Keywords: Coronary CT angiography; Revascularization; Decision-making
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
As the prospective, observational, cross-sectional study, the accuracy of CT angiography-based therapeutic decision-making for revascularization will be evaluated. The primary objective of this study is to evaluate the accuracy of CT angiography-based therapeutic decision-making for revascularization prior to conventional angiography whether CT angiography is an accurate non-invasive technique to determine the most appropriate therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 20 years old
* Patients who are scheduled for elective conventional coronary angiography and are undergone CT angiography prior to conventional coronary angiography.

Exclusion Criteria:

* Pregnant women or women with potential childbearing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited the tertiary hospital for coronary angiography who are undergone CT angiography prior to conventional coronary agniography
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy of CT angiography | 1day
  Sensitivity, specificity, positive predictive value, and negative predictive value for revascularization including PCI and CABG.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea